CLINICAL TRIAL: NCT06847945
Title: Changes of Acupoint Sensitization Characteristics on Gallbladder Meridian and Acupuncture Intervention Effect in Patients with Cervical Spondylosis
Brief Title: Observation on the Curative Effect of Acupuncture At Sensitized Points on Gallbladder Meridian in the Treatment of Neck Type Cervical Spondylopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LiChaoran (Other)
Responsible Party: Sponsor-Investigator, LiChaoran, Attending physician, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZSLL-KY-2023-040-03
Record Dates: First submitted 2025-02-14; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cervical Spondylopathy
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-meridian，non-acupoint group (Sham Comparator)
  Interventions: Procedure: Sham acupuncture
- Acupoint sensitization group (Experimental)
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Sham acupuncture — Patients in the non-meridian and non-acupoint group received sham acupuncture treatment at the position 2cm apart from the sensitized acupoint, once every other day for 30min each time, a total of 3 times for 1 week.
  Arms: Non-meridian，non-acupoint group
Procedure: Acupuncture — Patients in acupoint sensitization group were treated with pseudoacupuncture at the sensitized points once every other day for 30min each time, a total of 3 times for 1 week.
  Arms: Acupoint sensitization group

SUMMARY:
To investigate the changes of acupoint sensitization characteristics of patients with Neck Type Cervical Spondylopathy through Gallbladder meridian observe the curative effect of acupuncture intervention and optimize the clinical diagnosis and treatment plan of acupuncture treatment of Neck Type Cervical Spondylopathy

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria of Neck Type Cervical Spondylopathy.
* Age 18 to 65 years old gender is not limited.
* Clear awareness good compliance willing to cooperate with the study and accept the experimental arrangement.
* Physical examination may or may not be accompanied by positive signs of the musculoskeletal system (including limited motor function local tender points etc.).
* The visual analogue Scale (VAS) score was more than 3 points and less than 7 points (ranging from 0 to 10 points).
* Informed consent and sign informed consent.

Exclusion Criteria:

* It does not meet the diagnostic criteria and inclusion criteria of cervical spondylosis.
* Under 18 years of age or over 65 years of age;
* 2 weeks before the start of the experiment the relevant treatment of the disease or the use of relevant therapeutic drugs;
* Patients with other types of cervical spondylosis (cervical radiculopathy vertebral artery type cervical spondylosis cervical myelopathy sympathetic cervical spondylosis) or with other serious organic diseases and patients with neck and shoulder pain caused by non-neck diseases;
* Patients with cardiovascular and cerebrovascular liver kidney digestive system blood system and other serious life-threatening primary diseases or suffering from hemorrhagic diseases or skin diseases or pregnant or lactating women or have a history of cardiac pacemaker implantation;
* Previous history of neck surgery or neck fracture;
* Persons with confusion mental disorder or cognitive impairment;
* The skin at the test site has scars redness swelling heat and pain that affect the test result.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-05 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Before the start of treatment, immediately after the end of the third treatment, and four weeks after follow-up
  The visual Analogue Scale (VAS) ranging from 0 to 10, with higher scores reflecting more pain, stiffness and poorer physical function of the Cervical. Participants were asked to evaluate their current pain, and the pain nature was marked by X on the line above. 0 was classified as painless and 10 was classified as severe pain. The higher the score, the more obvious the pain.

SECONDARY OUTCOMES:
musculoskeletal ultrasound detection of cervical | Before the start of treatment, immediately after the end of the third treatment
Pressure pain threshold | Before the start of treatment, immediately after the end of the third treatment, and four weeks after follow-up
  The measurement result of FDX Force Gauge can quantify pain more objectively in clinical practice. And pressure pain threshold(PPT) at acupoints can be measured more objectively and accurately by FDX Force Gauge. The tester used a hand-held pain threshold test instrument to probe the acupoints.After switching on the machine, the comp peak mode was selected. The unit of measurement result is N.The figure on the display was zeroed before each measurement. The probe (1cm in diameter) was placed vertically on the acupoints of Gallbladder meridian. And the pressure was applied slowly and steadily at a constant speed(at a rate of 5N/s) downwards, and stopped immediately when the subject started to feel pain.The figure on the display is the pain threshold of the acupoint.Every acupoint was measured twice, with a 5-minute break between each measurement session.
The Neck Disability Index | Before the start of treatment, immediately after the end of the third treatment, and four weeks after follow-up
  The NDI consists of 10 items that cover various aspects of daily life affected by neck pain, including pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreational activities.Each item is scored on a scale from 0 to 5, where 0 indicates no disability and 5 represents the worst imaginable disability. The total score ranges from 0 to 50, which can also be expressed as a percentage by multiplying the raw score by 2.
  Interpretation of the scores is as follows:
  0-4: No disability 5-14: Mild disability 15-24: Moderate disability 25-34: Severe disability Over 34: Complete disability
Cervical range of motion scale | Before the start of treatment, immediately after the end of the third treatment, and four weeks after follow-up
  Subjects take a seated position, head in the middle, shoulders relaxed, both eyes looking straight ahead, forward flexion: normal flexion range of mition is between 35 °and 45 °; backward extension: the normal degree of backward extension is between 35 ° and 45 °; lateral flexion: normal lateral flexion range of mition is 45 °; rotate:the normal degree of rotation is between 60°and 80°. A range of motion instrument (Digital Angle Ruler)will be used to determine cervical spine movements. The device will be placed on the top or side of the head and the patient will be instructed to move the head as far as possible, without experiencing pain, in a standard fashion;right rotation, left rotation, flexion, extension, right lateral flexion and left lateral flexion. Within the range of cervical motion of patients, a larger value indicates a healthier cervical spine, while a smaller value indicates a more serious cervical mobility disorder.
The 12 items Short Form Health Survey | Before the start of treatment, immediately after the end of the third treatment, and four weeks after follow-up
  The 12-Item Short Form Health Survey (SF-12) is a widely used tool designed to assess overall health-related quality of life. It evaluates both physical and mental health domains through 12 questions, providing two composite scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).Scoring Range:Minimum Score: 0，Maximum Score: 100.Higher Scores: Indicate better health status. Higher PCS and MCS scores suggest better physical and mental well-being, respectively.Lower Scores: Indicate worse health status. Lower scores may suggest significant limitations in daily activities or poorer psychological well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Chaoran Li, Study Chair — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medicine University, Hangzhou, China

REFERENCES:
- [Derived] Li C, Wang J, Shao X, Wu Y, Qu X, Cai J, He L, Yu L, Xu R, Xia Y, Wang R, Zhang L, Qiu Y. Acupuncture at Sensitized Acupoints versus Sham Acupuncture for Neck-Type Cervical Spondylosis: Study Protocol for a Randomized Controlled Trial. J Pain Res. 2025 Dec 23;18:6963-6976. doi: 10.2147/JPR.S548317. eCollection 2025. PMID 41458188